CLINICAL TRIAL: NCT06501469
Title: Prospective, Observational Study to Identify Biomarkers in Parkinsonian Syndromes
Brief Title: Biomarkers in Parkinsonian Syndromes
Acronym: PROATYP
Status: Recruiting | Type: Observational
Sponsor: Non-profit organization for scientific research in Parkinson's disease and related disorders (Other)
Collaborators: Biomedical Research Foundation, Academy of Athens (Other)
Responsible Party: Sponsor
Other Study IDs: 642
Record Dates: First submitted 2024-06-20; First posted 2024-07-15 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease; Progressive Supranuclear Palsy; Multiple System Atrophy; Atypical Parkinsonism; Parkinsonism
Keywords: Parkinson's disease; Progressive Supranuclear Palsy; Multiple System Atrophy; Atypical Parkinsonism; Parkinsonism; Biomarkers
MeSH Terms: conditions — Parkinson Disease; Supranuclear Palsy, Progressive; Multiple System Atrophy; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational study to identify biomarkers in parkinson syndromes. Patients with parkinsonian syndromes at the early stages of disease will be recruited and will be followed up until their established clinical diagnosis or for at least 5 years. In this population, imaging and wet biomarkers as well as clinical data will b systematically collected.

ELIGIBILITY:
IΙnclusion Criteria:

* Written informed consent, including consent to monitoring
* Patients with Parkinsonism and disease duration < 2 years
* Patients with Parkinsonism and disease duration > 2 years
* Healthy individuals without any neurological disease

Exclusion Criteria:

* Drug-induced parkinsonism (eg, neuroleptics, lithium, valproic acid, metoclopramide).
* Metabolic conditions related parkinsonism (eg, Wilson's disease, hypoparathyroidism).
* Structural lesions on brain magnetic resonance imaging (MRI) that explain the symptoms, such as normal pressure hydrocephalus, moderate to severe chronic vascular encephalopathy, cerebral infarction, neoplasm
* Other serious diseases that indicate a life expectancy of <5 years.
* Active participation in other interventional clinical studies

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * patients with unclassified Parkinsonism and disease duration < 2 years
  * patients with suggestive, possible or probable progressive suprnanuclear palsy (PSP) and disease duration <2 years according to established clinical criteria
  * patients with possible, probable or clinically confirmed multiple system atrophy (MSA) and disease duration <2 years according to established clinical criteria
  * patients with parkinsonism (PD, MSA or PSP) and disease duration > 2 years according to established clinical criteria
  * patients with Parkinson's disease (PD) and disease duration < 2 years according to established clinical criteria
  * patients with Parkinson's disease (PD) and disease duration > 2 years according to established clinical criteria
  * healthy individuals without any neurological disease
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2029-03-25 (Estimated); Study Completion 2030-03-25 (Estimated)

PRIMARY OUTCOMES:
Demographics | At enrolment
  Age, gender, education, origin, race
Family history | At enrolment
  Family history of Parkinson's, dementia, tremor, other movement disorders, other neurological disorders
Age | At enrolment
  Age at onset in years
Disease duration | At enrolment
  Disease duration in years
First motor symptom | At enrolment
  First motor symptom time of onset
First non-motor symptom | At enrolment
  First non-motor symptom time of onset
Side of onset | At enrolment
  Side of onset of first motor symptom
Staging | At enrolment and every six months over 5 years
  Hoehn and Yahr stage (H&Y) stage (1-5, higher score indicate higher impairment)
Clinical scales - Unified Parkinson's disease rating scale (UPDRS) | At enrolment and every six months over 5 years
  Unified Parkinson's disease rating scale I-IV (UPDRS I-IV, 0-260; higher scores indicate higher impairment)
Clinical scales for Progressive supranuclear palsy (PSP) | At enrolment and every six months over 5 years
  Progressive supranuclear palsy rating scale (PSP-RS) (0-100; higher scores indicate higher impairment)
Clinical scales for Multiple system atrophy (MSA) | At enrolment and every six months over 5 years
  Unified Multiple system atrophy rating scale (UMSAPRS)(0-104; higher scores indicate higher impairment)
Clinical scales for PSP short | At enrolment and every six months over 5 years
  Progressive Supranuclear Palsy Clinical Deflicts Scale (PSP-CDS)(0-21; higher scores indicate higher impairment)
Clinical scales for apathy | At enrolment and every six months over 5 years
  Starkstein Apathy Scale (SAS) (0-56; higher scores indicate higher impairment)
Clinical scale for autonomic dysfunction | At enrolment and every six months over 5 years
  The Scale for Outcomes in Parkinson's disease for Autonomic symptoms - (0-100; higher scores indicate higher impairment)
Clinical scale for cognition | At enrolment and every six months over 5 years
  Montreal Cognitive Assessment (MOCA) (0-30, lower scores indicate higher impairment)
Clinical scale for frontal dysfunction | At enrolment and every six months over 5 years
  Frontal assessment battery (FAB) (0-18, lower scores indicate higher impairment)
Imaging outcome measures - nuclear medicine investigations | At enrolment
  (meta-iodobenzylguanidine) MIBG-Scintigraphy heart
Imaging outcome measures - Positron emission tomography (PET) | At enrolment
  fluorodeoxyglucose (FDG) -PET brain
Imaging outcome measures - Dopamine Transporters imaging (DaTScan) | At enrolment
  MRI brain
Imaging outcome measures - Magnetic resonance imaging (MRI) | At enrolment
  MRI brain
Blood samples analysis (DNA) | At enrolment
  Whole exome sequencing - genetic testing
Blood samples analysis (biomarkers, exosomes) | At enrolment and after 2 years
  Peripheral blood mononuclear cell (PBMCs), peripheral blood mononuclear cells, exosomes

CONTACTS AND LOCATIONS:
Overall Officials: Maria Stamelou, Prof Dr, Principal Investigator — HYGEIA Hospital
Locations (1):
- HYGEIA Hospital, Parkinson's disease and Movement Disorders Department, Athens, Greece